CLINICAL TRIAL: NCT04150783
Title: Computational Modeling of the Mature Unilateral Cleft Lip Nasal Deformity for Objective Assessment of Patient Nasal Function and Treatment Outcomes
Brief Title: Computational Modeling of Cleft Lip Nasal Deformity and Assessment of Nasal Function and Treatment Outcomes
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00102005; R01DE028554 (NIH)
Record Dates: First submitted 2019-10-24; First posted 2019-11-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cleft Lip and Nose; Nasal Obstruction
MeSH Terms: conditions — Cleft Lip; Nasal Obstruction | interventions — Wound Healing; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unilateral Cleft Lip Nasal Deformity (uCLND): uCLND patients who are scheduled to undergo surgical treatment for nasal obstruction as standard of care.
  Interventions: Procedure: Surgical repair for nasal obstruction
- Healthy Subjects: Existing data from healthy subjects with no prior symptoms of nasal obstruction used to create normative ranges for comparison to uCLND cohort.

INTERVENTIONS:
Procedure: Surgical repair for nasal obstruction — Patient reported quality of life questionnaires
  Other Names: observational, patient reported outcome measures
  Groups: Unilateral Cleft Lip Nasal Deformity (uCLND)

SUMMARY:
The purpose of this study is to use computers to simulate airflow in 3D construction of your nasal cavity generated from cone beam CT images. The results from computer simulations will help researchers identify the severity of cleft-induced nasal dysfunction and assess the impact of current treatment in restoring breathing function. The ultimate goal is to improve post-surgery outcomes to restore nasal breathing function to normal levels.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.
* Male or female, aged ≥18 years of age.
* Clinical diagnosis of unilateral cleft lip nasal deformity (uCLND)
* Scheduled to undergo elective surgery for nasal obstruction
* Scheduled to have a Cone Beam Computed Tomography (CBCT) as part of the pre- operative work-up for elective surgery.

Exclusion Criteria:

* Prior cleft rhinoplasty or septoplasty for correction of nasal obstruction
* Pregnant women: A pregnancy test will be performed within 48 hours of baseline
* Patients unable or unwilling to comply with study procedures outlined in protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral cleft lip nasal deformity scheduled to undergo elective surgery for nasal obstruction at the Duke Cleft and Craniofacial Center.
  Existing CBCT imaging data and QOL measures previously collected on healthy subjects will be used for comparison. Healthy subjects will not be prospectively enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Validation of computational fluid dynamics simulation with breathing measurement | 6 months
  Percent agreement between computational fluid dynamics simulated nasal resistance and nasal resistance from rhinomanometry breathing measurement
Validation of computational fluid dynamics simulation with in vitro experiment | 6 months
  Percent agreement between computational fluid dynamics simulated nasal resistance and nasal resistance measurement from in vitro experiment of 3D printed plastic nasal replica
Effectiveness of current surgery in restoring nasal function based on volumetric airflow | 6 months
  Analysis of significant difference in volumetric airflow rate between pre-surgery and post-surgery data from computational fluid dynamics simulations of patient-specific 3D nasal models generated from cone-beam computed tomography images.
Effectiveness of current surgery in restoring nasal function based on nasal resistance | 6 months
  Analysis of significant difference in nasal resistance between pre-surgery and post-surgery data from computational fluid dynamics simulations of patient-specific 3D nasal models generated from cone-beam computed tomography images
Effectiveness of current surgery in restoring nasal function based on nasal heat flux | 6 months
  Analysis of significant difference in nasal heat flux between pre-surgery and post-surgery data from computational fluid dynamics simulations of patient-specific 3D nasal models generated from cone-beam computed tomography images.
Effectiveness of current surgery in restoring nasal function based on nasal moisture flux | 6 months
  Analysis of significant difference in nasal moisture flux between pre-surgery and post-surgery data from computational fluid dynamics simulations of patient-specific 3D nasal models generated from cone-beam computed tomography images.
Anatomical sites of greatest nasal obstruction | 6 months
  Analysis on agreement of computational fluid dynamics identified anatomical sites of greatest nasal obstruction from pre-surgery 3D nasal models and actual surgical anatomical sites. CFD identified sites of greatest nasal obstruction are regions in the airway with highest nasal resistance.
Computational fluid dynamics based optimized treatment options for unilateral cleft lip nasal deformity patients based on volumetric airflow | 6 months
  Creation of virtual surgery nasal airway models based on computational fluid dynamics identified anatomical sites of greatest nasal obstruction. Computational fluid dynamics generated unilateral left and right side percent asymmetric will be computed used to identify the top three virtual surgery nasal airway models with best treatment potentials for unilateral cleft lip nasal deformity patients
Computational fluid dynamics based optimized treatment options for unilateral cleft lip nasal deformity patients based on nasal resistance | 6 months
  Creation of virtual surgery nasal airway models based on computational fluid dynamics identified anatomical sites of greatest nasal obstruction. Computed nasal resistance will be used to identify the top three virtual surgery nasal airway models with best treatment potentials for unilateral cleft lip nasal deformity patients
Computational fluid dynamics based optimized treatment options for unilateral cleft lip nasal deformity patients based on nasal heat flux | 6 months
  Creation of virtual surgery nasal airway models based on computational fluid dynamics identified anatomical sites of greatest nasal obstruction. Computed nasal moisture flux will be used to identify the top three virtual surgery nasal airway models with best treatment potentials for unilateral cleft lip nasal deformity patients

SECONDARY OUTCOMES:
Change in patient-reported outcome (PRO) measures | baseline, 2 weeks, 8 weeks, 6 months, 12 months
  Change PRO measures as measured by NOSE questionnaire
Change in patient-reported outcome (PRO) measures | baseline, 2 weeks, 8 weeks, 6 months, 12 months
  Change PRO measures as measured by SCHNOS questionnaire
Change in patient-reported outcome (PRO) measures | baseline, 2 weeks, 8 weeks, 6 months, 12 months
  Change PRO measures as measured by CLEFT-Q questionnaire
in vitro analysis for top three virtual surgery nasal models with best treatment based on nasal pressure | 6 months
  in vitro analysis from 3D printed plastic nasal replica of top three virtual surgery nasal models with best treatment potential will be done using unilateral airflow pressure.
in vitro analysis for top three virtual surgery nasal models with best treatment based on unilateral volumetric airflow | 6 months
  in vitro analysis from 3D printed plastic nasal replica of top three virtual surgery nasal models with best treatment potential will be done using unilateral volumetric airflow rate.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Frank-Ito, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center and affiliated practices, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Russel SM, Chiang H, Finlay JB, Shah R, Marcus JR, Jang DW, Abi Hachem R, Goldstein BJ, Frank-Ito DO. Characterizing Olfactory Dysfunction in Patients with Unilateral Cleft Lip Nasal Deformities. Facial Plast Surg Aesthet Med. 2023 Nov-Dec;25(6):457-465. doi: 10.1089/fpsam.2022.0367. Epub 2023 May 2. PMID 37130297